CLINICAL TRIAL: NCT01791608
Title: Effect of Zinc Sulphate and Zinc Amino Acid Chelate in Prevention Acute Diarrhea and Acute Respiratory Infection, Medellín 2012
Brief Title: Zinc Sulphate vs. Zinc Amino Acid Chelate
Acronym: ZAZO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CES University (Other)
Collaborators: Nutreva S.A.S. (Unknown); Foundation Child Care - FAN (Other)
Responsible Party: Principal Investigator, Juliana Sanchez,MG, Principal investigator, CES University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ZAZO-01
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Diarrhea; Acute Respiratory Infection
Keywords: Child, Preschool; Dietary Zinc; Zinc sulfate; zinc-glycine chelate
MeSH Terms: conditions — Diarrhea | interventions — Zinc Sulfate; Dietary Supplements; Milk; Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Zinc sulphate (Active Comparator): Preschool children healthy enrolled in FAN Foundation of Medellin, which will be supplied with zinc sulphate
  Interventions: Dietary Supplement: Zinc sulfate as dietary supplementation
- Zinc Amino Acid Chelate (Experimental): Preschool children healthy enrolled in FAN Foundation of Medellin , which will be supplied with zinc amino acid chelate
  Interventions: Dietary Supplement: Zinc amino acid chelate as dietary supplementation
- Milk without fortification (Placebo Comparator): Milk without zinc
  Interventions: Dietary Supplement: Milk without fortification without zinc

INTERVENTIONS:
Dietary Supplement: Zinc sulfate as dietary supplementation — Zinc sulfate as dietary supplementation
  Arms: Zinc sulphate
Dietary Supplement: Zinc amino acid chelate as dietary supplementation — Zinc amino acid chelate as dietary supplementation
  Arms: Zinc Amino Acid Chelate
Dietary Supplement: Milk without fortification without zinc — Milk without fortification
  Other Names: Milk without zinc
  Arms: Milk without fortification

SUMMARY:
Acute respiratory infection and acute diarrhea are among the most prevalent diseases of childhood increase the burden of morbidity and mortality in children under 5 years.

Among the possible strategies for its prevention is important to count on good nutritional status for use in developing a good immune response to infections. Zinc deficiency has been shown to favor the development of infections and has been considered a real public health problem.

Within the zinc compounds used are zinc amino acid chelate and zinc sulphate, the first that has shown evidence of being better absorbed and tolerated.

We propose a study showing the effectiveness of zinc amino acid chelate and zinc sulphate in the prevention of acute diarrheal disease and acute respiratory infection.

ELIGIBILITY:
Inclusion Criteria:

Children who

* Belong to institute FAN in Medellín
* Attend full time to institute FAN (eight hours)
* Have 2 to 5 years

Exclusion Criteria:

Children who

* Children at the began of the study are with acute diarrheal disease and acute respiratory infection.
* Recurrent pneumonia, cystic fibrosis, gastrointestinal malformations, persistent diarrhea of any cause, inflammatory bowel disease.
* Failure to attend the educational institution for more than 10 days
* No consumption of zinc supplementation for more than 10 days, because of insistence to the school

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Incidence acute diarrheal disease and acute respiratory infection | Up to 16 weeks
  Preschool children will drink fortified milk with zinc amino acid chelate, zinc sulfate or milk without fortification. Fortnightly monitoring will be investigating the presence of infection (acute diarrheal disease and respiratory infections). Supervision and monitoring will be carried out for four months.

SECONDARY OUTCOMES:
Adverse reaction | Fortnightly. During 4 months of intervention
  The caregiver recorded daily if the child had an adverse reaction such as abdominal pain, nausea and vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Liliana LM Montoya, Master, Study Director — CES University
Locations (1):
- CES University, Medellín, Antioquia, Colombia

REFERENCES:
- [Derived] Sanchez J, Villada OA, Rojas ML, Montoya L, Diaz A, Vargas C, Chica J, Herrera AA. [Effect of zinc amino acid chelate and zinc sulfate in the incidence of respiratory infection and diarrhea among preschool children in child daycare centers]. Biomedica. 2014 Jan-Mar;34(1):79-91. doi: 10.1590/S0120-41572014000100011. Spanish. PMID 24967861